CLINICAL TRIAL: NCT02584322
Title: Fast Tracking in VATS Lobectomy: A Prospective, Historically Controlled, Propensity-Matched Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14.386
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ERAS patients (Experimental): Enhanced recovery pathway
  Interventions: Other: Enhanced Recovery pathway

INTERVENTIONS:
Other: Enhanced Recovery pathway — The enhanced recovery pathway consists of postoperative medical orders including nursing care, investigations and tests, and other peri-operative orders. The enhanced recovery pathway is standardized for all patients, and can be discontinued at any time when clinical judgment mandates (i.e. patient has a severe complication).

SUMMARY:
Currently, at the CHUM - Notre-Dame Hospital, there is no standardized patient care pathway for patients undergoing Video Assisted Thoracic Surgery (VATS) lobectomy. The investigators goal is to implement an Enhanced Recovery Program (ERP) for patient undergoing VATS lobectomy.

The care given to patient prior to the implementation of this protocol was different amongst patients and depended on the surgeon's preferences. The implementation of this ERP will permit a reproducible and routine management for patients following their surgery.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer related death in men and women worldwide annually. In North America in 2009, an estimated 246,000 people were diagnosed with lung cancer, and 178,000 died as a result. Lobectomy consists of the surgical removal of an anatomic lobe of the lung. It represents the standard of care in the treatment of malignant lesions involving one lobe of the lung. This operation can be performed either with a chest incision with rib spreading (thoracotomy) or with a minimally invasive approach which does not include rib spreading (thoracoscopy - Video Assisted Thoracoscopic Surgery; VATS).

In the last decade, the trend towards implementation of protocols to enhance patient recovery and diminish length of stay has been gaining popularity and increasing in prevalence. Those protocols are commonly referred to as fast track surgery or enhanced recovery after surgery protocol. The rationale behind these protocols is that by combining multimodal therapies that reduce surgical stress, having good pain control post-operatively, and involving the patient in this process, the treating team has the potential to reduce length of stay.

In the last few years, many surgeons in their respective centers have implemented the use of fast track surgery in the thoracic surgery service. It has been shown to be a safe and effective method for managing postoperative patients after lobectomy. Fast track surgery is a systemic approach to the management of surgical patients, where all the different actions to take postoperatively are standardized and reproducible. Fast track surgery has the potential to diminish the rate of postoperative complications, the length of stay, and achieve a similar patient recovery. In an era, where medical costs are on the rise, hospital beds are limited and nursing staff not always available, fast track surgery has the potential to improve increase throughput, improve efficiency, decrease costs and improve surgical productivity.

Currently, at the CHUM - Notre-Dame Hospital, there is no standardized patient care pathway for patients undergoing VATS lobectomy. The care given to patient prior to the implementation of this protocol was different amongst patients and depended on the surgeon's preferences. The implementation of this Enhanced Recovery Program (ERP) will permit a reproducible and routine management for patients following their surgery.

The principal outcomes that will be compared amongst patients pre and post implementation of this protocol will be the length of stay and the number of complications. The investigators think that the results will be different between these two groups. The rational for this is due to the fact that the patients in this Enhanced Recovery Program will have: (1) their urinary catheter removed sooner, (2) their thoracic drain removed earlier and (3) they will be mobilized more quickly. These differences will enable these patients to potentially have less complications post operatively and decrease their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a VATS lobectomy

Exclusion Criteria:

* Less than 18 year old, inability to consent, VATS lobectomy conversion to open lobectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 30 days post operative
  Number and Severity of Complications

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Montreal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Howington JA, Gunnarsson CL, Maddaus MA, McKenna RJ, Meyers BF, Miller D, Moore M, Rizzo JA, Swanson S. In-hospital clinical and economic consequences of pulmonary wedge resections for cancer using video-assisted thoracoscopic techniques vs traditional open resections: a retrospective database analysis. Chest. 2012 Feb;141(2):429-435. doi: 10.1378/chest.10-3013. Epub 2011 Jul 21. PMID 21778260
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Carrott PW Jr, Jones DR. Teaching video-assisted thoracic surgery (VATS) lobectomy. J Thorac Dis. 2013 Aug;5 Suppl 3(Suppl 3):S207-11. doi: 10.3978/j.issn.2072-1439.2013.07.31. PMID 24040525
- [Background] Flores RM, Park BJ, Dycoco J, Aronova A, Hirth Y, Rizk NP, Bains M, Downey RJ, Rusch VW. Lobectomy by video-assisted thoracic surgery (VATS) versus thoracotomy for lung cancer. J Thorac Cardiovasc Surg. 2009 Jul;138(1):11-8. doi: 10.1016/j.jtcvs.2009.03.030. PMID 19577048
- [Background] McKenna RJ Jr, Mahtabifard A, Pickens A, Kusuanco D, Fuller CB. Fast-tracking after video-assisted thoracoscopic surgery lobectomy, segmentectomy, and pneumonectomy. Ann Thorac Surg. 2007 Nov;84(5):1663-7; discussion 1667-8. doi: 10.1016/j.athoracsur.2007.05.058. PMID 17954081
- [Background] Zehr KJ, Dawson PB, Yang SC, Heitmiller RF. Standardized clinical care pathways for major thoracic cases reduce hospital costs. Ann Thorac Surg. 1998 Sep;66(3):914-9. doi: 10.1016/s0003-4975(98)00662-6. PMID 9768951
- [Background] Cerfolio RJ, Pickens A, Bass C, Katholi C. Fast-tracking pulmonary resections. J Thorac Cardiovasc Surg. 2001 Aug;122(2):318-24. doi: 10.1067/mtc.2001.114352. PMID 11479505
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278